CLINICAL TRIAL: NCT03734250
Title: The Effect of D Vitamin Status on Different Neuromuscular Blocker Agents Reverse Time
Brief Title: D Vitamin Effects on Neuromuscular Blocker Reverse Time
Status: Completed | Type: Observational
Sponsor: Duzce University (Other)
Responsible Party: Sponsor
Other Study IDs: 2014.04.02.221
Record Dates: First submitted 2018-10-06; First posted 2018-11-07 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Vitamin D Deficiency; Neuromuscular Block; Neuromuscular Block Problem
Keywords: Sugammadex; Neostigmine; Anesthesia; Neuromuscular blockers; Reverse time; Vitamin D
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Venous blood samples 20 ml
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group Sugammadex HD: Sugammadex used as neuromuscular blocker reverse agent with Vitamin D status equal or above 30ng/ml
- Group neostigmine HD: Neostigmine used as neuromuscular blocker reverse agent with Vitamin D status equal or above 30 ng/ml
- Group Sugammadex LD: Sugammadex used as neuromuscular reverse agent with Vitamin D status under 30 ng/ml
- Group Neostigmine LD: Neostigmine used as neuromuscular reverse agent with Vitamin D status under 30ng/ml

SUMMARY:
Background/aim: Investigators aimed to investigate the effect of D vitamin levels on Sugammadex and Neostigmine reverse durations in the study.

Materials and methods: Eighty patients between 18 and 65 years, with ASA I-III status who were undergoing surgery under general anaesthesia were included the study. All patients were randomly divided into two groups with double blindness and 1.25 (OH) 2 vitamin D, 25 (OH) 2 vitamin D, and calcium levels were measured. At the end of the operation, 2 mg/kg of Sugammadex was administered to one group and Atropine + Neostigmine to the other group. The patients were also divided into two groups as to whether their vitamin D levels were ≥ 30 ng/mL or below.

A train of four values was recorded after a hypnotic agent was given at the beginning and throughout the operation. The time to complete the disappearance of response to TOF stimulation was recorded as T0.

End of the operation: When 2 responses to TOF stimulation were taken, the following times were recorded until the extubation phase by administering at least 2 mg/kg of Sugammadex or 0.05 mg/kg of Neostigmine 0.05 mg/kg of Atropine per kg of body weight. The time until the TOF value reached 50,70,90% and extubation were recorded.

DETAILED DESCRIPTION:
Prospective observational study was carried out in the same centre after the approval of the University Hospital by the ethical committee of non-invasive research (Duzce University, School of Medicine, Ethics Committee of Non-invasive clinical research approval for application Date: 11.10.2013, Decision Number: 2013/439) and done by Anaesthesiology Department in the same centre. This research was also funded by our University Scientific Research Project Coordinating Department (2014.04.02.221).

Eighty-four patients with ASA I-III status, undergoing surgery under general anaesthesia between the ages of 18 and 65 years were included the study. Twenty millilitre blood samples were taken from the antecubital ven before the operation, after taken the approval of all patients. 1.25 (OH) 2 vitamin D, 25 (OH) 2 vitamin D, calcium, magnesium, phosphorus and parathormone levels were measured in the blood samples. All patients were randomly divided into two groups with double blindness. At the end of the operation, a 2 mg/kg dose of Sugammadex (Group Sugammadex n = 40) and 0.55 mg/kg + 0.015 mg/kg atropine Neostigmine (to the other group) were administered intravenously. The patients were also divided into two groups, having vitamin D levels above 30 ng/mL and below 30 ng/mL.

All patients were connected to a kinemyograph, which placed the neuromuscular transmission (NMT) module (GE Health Care) on the patients' adductor pollicis muscle before the anaesthesia induction. Patients body temperature were monitored and maintained within 35-37 0 C. Subsequently, the hypnotic agent was given at the beginning of the operation and Train of Four (TOF) values were recorded as % values throughout the operation. All patients received 2 mg of Midazolam intravenously for premedication. All patients were monitored by standard monitoring and received 2 mg / kg Propofol and 1 mcg/kg Fentanyl. Train of Four (TOF) stimulation started at 1 Hz intervals at a frequency of 2 Hz in 1-minute intervals. The initial values determined were recorded as the baseline TOF values and 0.5 mg / kg Rocuronium (Esmeron amp, Organon, Holland) was administered intravenously, which was calculated on ideal body weight. The time to complete disappearance of response to TOF stimulation was recorded as T0 and endotracheal intubation was performed.

Anaesthetic maintenance was proven by 50% oxygen + 50% air + 2% volume Sevoflurane via endotracheal tube. Remifentanil was administered intravenously at 0.05-1 mcgr /kg /h. When a 2-point response to TOF was received, the muscle relaxant was administered in repeated doses as 10 mg of Rocuronium.

The total muscle relaxant quantities were recorded. At the end of the operation: when 2 responses to TOF stimulation were taken, the following times were recorded until the extubation phase by administering at least 2 mg/kg of Sugammadex (Bridion flk, Merck Sharp & Dohme) or 0.05 mg/kg of Neostigmine (Neostigmin amp, Adeka, Turkey) and 0.05 mg/kg of Atropine per kg body weight.

T0.5: The time until the TOF value reached 50% T0.7: The time until the TOF value reached 70% T0.9: The time until the TOF value reached 90% Teks: Time to extubation.

Patients, who were able to open their eyes with spontaneous breathing, had a tidal volume of 10 ml/kg, according to ideal body weight during spontaneous breathing, pulse oximetry values above 95%, headache for 5 seconds, and TOF values above 90%.

Statistical analysis

Investigators used the independent samples t-test for two variables, continuous variables for comparison, and the Pearson Chi-square test for categorical variables. Repeated measures ANOVA was used to examine the interaction between drug groups and TOF measurement time. Co-effects of drug groups and vitamin D subgroups were examined by two-way analysis of variance (ANOVA). Repeated measures ANOVA, one of the three-factor differentials, were used to examine the TOF measurement time interaction of drug effects and vitamin D subgroups' concerted effects. Statistical analyses were performed with the SPSS v.22 packet program and the significance level was taken as 0.05.

ELIGIBILITY:
Inclusion:

* undergoing surgery under general anesthesia
* ASA I-III
* between the ages of 18 and 65 years old.

Exclusion

* diabetes
* kidney
* muscle
* hepatic diseases
* metabolic diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eighty four patients with ASA I-III status undergoing surgery under general anesthesia between the ages of 18 and 65 years were included the study
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Reverse times | 10 minute
  The time until the TOF value reaches 50,70,90% and extubation were recorded.

SECONDARY OUTCOMES:
Rocuronium effect unset time | 4 minute
  Time to complete disappearance of response to TOF stimulation was recorded as T0

CONTACTS AND LOCATIONS:
Overall Officials: İlknur S Yorulmaz, Dr, Principal Investigator — Duzce University

REFERENCES:
- [Background] Holick MF. Vitamin D status: measurement, interpretation, and clinical application. Ann Epidemiol. 2009 Feb;19(2):73-8. doi: 10.1016/j.annepidem.2007.12.001. Epub 2008 Mar 10. PMID 18329892
- See also: Pubmed — https://www.ncbi.nlm.nih.gov/pubmed/18329892